CLINICAL TRIAL: NCT04593056
Title: Replication of the ROCKET-AF Anticoagulant Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-ROCKET-AF
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Warfarin; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Warfarin: Reference group
  Interventions: Drug: Warfarin
- Rivaroxaban: Exposure group
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Warfarin — Warfarin dispensing claim is used as the reference
  Groups: Warfarin
Drug: Rivaroxaban — Rivaroxaban dispensing claim is used as the exposure
  Groups: Rivaroxaban

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Please see: https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates: Market availability of rivaroxaban in the U.S. started on November 4, 2011. For Marketscan: November 4, 2011 -Dec 31, 2018 (end of data availability). For Optum: November 4, 2011 -Dec 31, 2019 (end of data availability). For Medicare: November 4, 2011 -Dec 31, 2017 (end of data availability)

Inclusion Criteria:

* 1. Patients 18 years of age or older
* 2. Non-valvular atrial fibrillation
* 3. Non-valvular atrial fibrillation 14 days or after the previous diagnosis of AF in inclusion 2
* 4. History of prior ischemic stroke, TIA, systemic embolism or two or more of the following risk factors:

  * 4a. Heart failure and/or left ventricular ejection fraction ≤35%
  * 4b. Hypertension (defined as use of antihypertensive medications within 6 months before the screening visit or persistent systolic blood pressure above 140 mmHg or diastolic blood pressure above 90 mmHg)
  * 4c. Patients 75 years of age or older
  * 4d. Diabetes mellitus (defined as a history of type 1 or type 2 diabetes mellitus or use of antidiabetic medications within 6 months before screening visit)

Exclusion Criteria:

* 1. Cardiac-related conditions

  * 1a. Hemodynamically significant mitral valve stenosis
  * 1b. Prosthetic heart valve (annuloplasty with or without prosthetic ring, commissurotomy and/or valvuloplasty are permitted)
  * 1e. Known presence of atrial myxoma or left ventricular thrombus
  * 1f. Active endocarditis
* 2. Hemorrhage-related risk criteria

  * 2a. Active internal bleeding
  * 2b. History of or condition associated with increased bleeding risk including, but not limited to:

    * Major surgical procedure or trauma within 30 days before the randomization visit
    * Clinically significant gastrointestinal bleeding within 6 months before the randomization visit
    * History of intracranial, intraocular, spinal, or atraumatic intra-articular bleeding
    * Chronic hemorrhagic disorder
    * Known intracranial neoplasm, arteriovenous malformation, or aneurysm
  * 2d. Platelet count < <90,000/μL at the screening visit
  * 2e. Sustained uncontrolled hypertension: systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100
* 3. Concomitant conditions and therapies

  * 3a. Severe, disabling stroke (modified Rankin score of 4 to 5, inclusive) within 3 months or any stroke within 14 days before the randomization visit
  * 3b. Transient ischemic attack within 3 days before the randomization visit
  * 3c. Indication for anticoagulant therapy for a condition other than atrial fibrillation (e.g., VTE)
  * 3d. Treatment with:

    * Aspirin >100 mg daily
    * Aspirin in combination with thienopyridines within 5 days before randomization
    * Intravenous antiplatelets within 5 days before randomization
    * Fibrinolytics within 10 days before randomization
    * Note: Aspirin ≤100 mg monotherapy is allowed and thienopyridine monotherapy is allowed.
  * 3f. Systemic treatment with a strong inhibitor of cytochrome P450 3A4, such as ketoconazole or protease inhibitors, within 4 days before randomization, or planned treatment during the time period of the study
  * 3g. Treatment with a strong inducer of cytochrome P450 3A4, such as rifampin/rifampicin, within 4 days before randomization, or planned treatment during the time period of the study
  * 3h. Anemia (hemoglobin <10 g/dL) at the screening visit
  * 3i. Pregnancy or breast-feeding
  * 3k. Known HIV infection at time of screening
  * 3l. Calculated CLCR <30 mL/min at the screening visit (refer to Attachment 4 for calculating CLCR)
  * 3m. Known significant liver disease (e.g., acute clinical hepatitis, chronic active hepatitis, cirrhosis), or ALT >3 x the ULN
* 4. Study participation and follow-up-related criteria

  * 4a. Serious concomitant illness associated with a life expectancy of less than 2 years
  * 4b. Drug addiction or alcohol abuse within 3 years before the randomization visit
  * 4f. Inability or unwillingness to comply with study-related procedures

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will involve a new user, parallel group, cohort study design comparing rivaroxaban to warfarin. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of rivaroxaban or the comparator drug (cohort entry date). Follow-up for the outcome, begins the day after drug initiation.
Sampling Method: Probability Sample
Enrollment: 102636 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
Relative hazard of composite outcome of Stroke and Systemic Embolism | [Time Frame: Through study completion (a median of 98-119 days)]
  Relative hazard of composite outcome of Stroke and Systemic Embolism - Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham And Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT04593056/Prot_SAP_001.pdf